CLINICAL TRIAL: NCT05079386
Title: Early Clinical Feasibility Study of a New Voice Prosthesis
Brief Title: Clinical Feasibility of a New Voice Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: N21VEG
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Laryngectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- New Voice Prosthesis (Experimental): Patients will use the New Voice Prosthesis for two weeks to investigate short term feasibility and explore limitations and advantages. If the patient wishes to leave the New Voice Prosthesis in situ, this will be allowed under the condition that the subject agrees to remain in the study and report (adverse) events on an ongoing basis, until the device is removed after a maximum of 12 months.
  Interventions: Device: New Voice Prosthesis

INTERVENTIONS:
Device: New Voice Prosthesis — Replacement of the current prosthesis with the experimental device and use the New Voice Prosthesis for the duration of two weeks with the option of leaving the device in situ until replaced for device failure or other reason, with a maximum of 12 months.

SUMMARY:
The objective of this clinical investigation is to evaluate the short-term clinical feasibility of a new voice prosthesis and explore its acceptability, limitations and advantages. As a result of the evaluations, design changes may be implemented and evaluated until the optimal design has been determined, or until it is decided not to pursue further development of the device. Main outcome will be the patient's acceptance of the voice prosthesis, secondary outcomes are stickiness of the valve mechanism and speech.

ELIGIBILITY:
Inclusion Criteria:

* Laryngectomized patients using either the Provox Vega 22.5 or the Provox ActiValve Light voice prosthesis, with a length of 4, 6, 8, or 10 mm
* 18 years and older

Exclusion Criteria:

* Current tracheoesophageal puncture problems such as enlarged puncture or infection
* Active recurrent or metastatic disease (medical deterioration)
* The use of ActiValve Strong/XtraStrong or XtraSeal
* Unable to understand the Patient Information and/or unable to give Informed Consent
* The previous 2 VPs had a device lifetime > 12 months
* History of oral resections negatively affecting speech

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Patient acceptability | 2 week
  Patient recorded acceptability of the voice prosthesis based on study specific questionnaires covering: 1) Experienced stickiness, 2) Effort to speak and 3) maintenance of voice prosthesis. Assessed by Yes/No and multiple choice questions.

SECONDARY OUTCOMES:
Voice Assessment - Maximum phonation | Baseline and 2 weeks
  Longest maximum phonation time in seconds out of 2 consecutive attempts. Assessed with current Voice prosthesis and the New Voice Prosthesis.
Voice Assessment - Highest volume | Baseline and 2 weeks
  Highest volume in hertz. Assessed with current Voice prosthesis and the New Voice Prosthesis.
Voice Assessment - Lowest Volume | Baseline and 2 weeks
  Lowest volume in hertz. Assessed with current Voice prosthesis and the New Voice Prosthesis.
Voice Assessment - Softness | Baseline and 2 weeks
  Speaking as soft as possible in decibels. Assessed with current Voice prosthesis and the New Voice Prosthesis.
Voice Assessment - Loudness | Baseline and 2 weeks
  Speaking as loud as possible in decibels. Assessed with current Voice prosthesis and the New Voice Prosthesis.
Voice Assessment - Glide tones | Baseline and 2 weeks
  Successful completion of glide town, from low to high. Assessed with current Voice Prosthesis and the New Voice Prosthesis.
Quality of Life by EQ-5D-5L | Baseline and 2 weeks
  Patient reported, the descriptive system assesses health in five dimensions, from which a health state index score is calculated, range from 0 to 1, with higher scores indicating higher health utility
Voice Handicap Index - 10 | Baseline and 2 weeks
  Validated tool to assess Voice handicap. Statements on participant's voice quality and effect on social life are assessed by a five-point Likert-scale, ranged from 0-4, with high scores indicating more handicap (0 = Never, 4 = Always).
Device life | Baseline, and week 52
  Device life of two previous Voice prosthesis and device life of the New Voice Prosthesis in the long-term part of study.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel van den Brekel, Prof, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute: NKI, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heirman AN, Tellman RS, van der Molen L, van Son R, van Sluis K, Halmos GB, Van den Brekel MWM, Dirven R. The acceptance and voice quality of a new voice prosthesis 'Vega High performance' - a feasibility study. Acta Otolaryngol. 2023 Aug;143(8):721-729. doi: 10.1080/00016489.2023.2241876. Epub 2023 Sep 1. PMID 37656679